CLINICAL TRIAL: NCT07297615
Title: Accuracy of Individualized 3D Reconstruction in Predicting Liver Resection Volume: A Prospective Study
Brief Title: 3D Liver Volumetry
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1465/2025
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Liver Surgery; Liver Cancer; Surgical Planning; Liver; Volumetric Analysis; 3D-reconstruction
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volumetry through 3D reconstruction (Experimental): Preoperative liver volumetry using individualized 3D reconstructions to guide major hepatectomy, optimize resection planning, and improve prediction of the future liver remnant.
  Interventions: Diagnostic Test: 3d reconstruction

INTERVENTIONS:
Diagnostic Test: 3d reconstruction — Preoperatively, every patient in this study will undergo an individualized 3D reconstruction of their liver to perform accurate volumetry.

SUMMARY:
The study aims to improve preoperative evaluation of liver resection volume in patients undergoing major hepatectomies. Accurate prediction of the planned resection and the future liver remnant (FLR) is critical to minimize the risk of postoperative liver failure, which is associated with increased morbidity and mortality. Conventional imaging-based volumetry may have limited accuracy. This study investigates the use of individualized 3D liver models combined to enhance visualization and volumetric analysis of liver anatomy and resection boundaries.

Patients are recruited in the liver outpatient clinic and, upon consent, preoperative 3D models are created using Medics 3D. During surgery, the planned resection is guided by the individualized 3D models. Postoperatively, the resected specimen undergoes CT-based volumetry to compare the predicted resection volume from the 3D model with the actual volume. Routine postoperative follow-up is conducted. The study aims to optimize surgical planning, enhance the accuracy of future liver remnant prediction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) undergoing open or minimally invasive major liver resection at the Clinical Division of General, Visceral and Transplant Surgery who provide written informed consent prior to participation will be included.

Exclusion Criteria:

* Patients unable to provide informed consent will be excluded.
* Minor resections.
* Contraindications to MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the preoperative volumetry of the liver portion planned for resection using a 3D model and comparison with the postoperative resection specimen volume. | Approximately 2-3 weeks are required between preoperative volumetry and postoperative volumetry comparison.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz - Department of Surgery, Division of General, Visceral and Transplantationsurgery, Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No